CLINICAL TRIAL: NCT05684861
Title: Serum TWEAK Levels in Acne Vulgaris Patients Treated With Oral Isotretinoin
Brief Title: Serum TWEAK Levels in Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Hassan Mohammed Ibrahim, Associate professor, South Valley University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: SVU MED DVA021 4 22 11 508
Record Dates: First submitted 2023-01-01; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I patients (Active Comparator): 90 patients with acne vulgaris Patients classified according to the global acne grading system(GAGS) into moderate, severe, and very severe cases
  Interventions: Drug: Isotretinoin; Diagnostic Test: ELISA Assays of Serum TWEAK.
- Control group (Active Comparator): 60 age-sex-matched healthy subjects as a control group
  Interventions: Diagnostic Test: ELISA Assays of Serum TWEAK.

INTERVENTIONS:
Drug: Isotretinoin — systemic isotretinoin was given to all 90 patients , dose was prescribed according to weight for 3 months
  Arms: Group I patients
Diagnostic Test: ELISA Assays of Serum TWEAK. — : From each subject, 5mL of blood was collected into vacutainers before and after treatment with isotretinoin. The blood samples were centrifuged at 3000g for 10 min at a temperature of 4°C, then . Quantitative determinations for serum TWEAK were achieved using the corresponding commercially available ELISA kit supplied by the AssayMax

SUMMARY:
Evaluate the serum level of TWEAK in patients with AV and their relations before and after treatment with isotretinoin.

DETAILED DESCRIPTION:
Acne vulgaris is a chronic inflammatory disease of the pilosebaceous follicles, characterized by comedones, papules, pustules, cysts, nodules, and occasionally scars. Its pathogenesis includes follicular hyperkeratinization, sebaceous hypersecretion due to androgen stimulation, follicular colonization by Propionibacterium acnes, immune and inflammatory responses. It affects the face, anterior chest, and upper back . Inflammation is regarded as a key component in the pathogenesis of acne . An increase in the activity of the pro inflammatory cytokine, interleukin (IL) 1, is observed before the beginning of hyperproliferation around the uninvolved follicles and is thought to trigger the activation of keratinocyte proliferation. Nuclear factor kappa beta (NF κβ) regulated mRNA gene levels of the cytokines tumour necrosis factor (TNF) α, IL 1 β, IL 8 and IL 10 levels also affected.

Isotretinoin (13-cis retinoic acid) is a synthetic analog of vitamin A. Its oral form is prescribed for severe cases which are resistant to other treatments.

Tumor necrosis factor (TNF)-like weak inducer of apoptosis (TWEAK) belongs to the TNF superfamily. It has an important role in the regulation of cell growth, apoptosis, angiogenesis, and immune reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified according to the global acne grading system(GAGS) into moderate, severe, and very severe cases

Exclusion Criteria:

* Pregnant and lactating women, patients with renal, GIT, skeletal, psychiatric, and endocrine disorders, sarcoidosis, and patients receiving drugs such as diuretics, multivitamins, anticonvulsants, glucocorticoids, erythromycin, estrogen compound pill were excluded.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
serum level of TWEAK | 12 weeks
  To evaluate the serum level of TWEAK in patients with moderate to severe acne vulgaris.

SECONDARY OUTCOMES:
evaluate the effect of systemic isotretinoin on serum TWEAK level | 12 weeks
  the comparison of the serum TWEAK before and after treatment with isotretinoin in moderate and severe cases of acne vulgaris.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Ibrahim, professor, Study Director — South Valley University
Locations (1):
- South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No